CLINICAL TRIAL: NCT03019952
Title: Effectiveness of the Care Coordination, Assessment, and Responsive Engagement Program for Transition-aged Adolescents (t-CARE) With ASD
Acronym: t-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Pennsylvania Bureau of Autism Services (Other)
Responsible Party: Principal Investigator, Michael Murray, Associate Professor of Psychiatry, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00003849
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Care Coordination Visit — This is a longitudinal study. Adolescents or young adults with autism will participate in this study. Participants will be required to complete a baseline of assessment measures at enrollment and then monthly assessments (described in the study procedures below) during the first (approximately) 10-15 minutes of each visit with the t-CARE coordinator. The remainder of the visit will focus on care coordination and clinical treatment goals.

SUMMARY:
An analysis of data for adolescents and young adults diagnosed with Autism Spectrum Disorders (ASDs) who are evaluated as part of the Care Coordination, Assessment, and Responsive Engagement for transition-aged adolescents (t-CARE) program which replaced the former Autism Life Care Model (ALCM), which was a clinical program implemented between Fall 2014 and April 2016. The individuals enrolled in the program will be administered a standardized assessment battery during each visit with the care coordinator or study coordinator. The proposed study will analyze data gathered during each of the assessment periods in order to check the efficacy and viability of the protocol.

DETAILED DESCRIPTION:
Current collaboration between individuals, families, and providers through in-person meetings are extremely infrequent, costly, and occur most often when providers are intimately involved as part of a multidisciplinary team in a single setting such as at a school. Often, little information is transmitted between providers and/or school personnel in determining treatment goals and interventions. Furthermore, the transmission of information is often provider to provider or school personnel to provider, which excludes direct patient-input and lessens transparency in decision making. In an effort to improve current care and therefore improve successful adult transitions for adolescents with ASD, t-CARE is designed to mimic multidisciplinary team meetings. These meetings are incredibly impactful as they include direct individual and family involvement through facilitated information-sharing, while also maintaining patient-centered care across multiple providers and complex systems of care.

ELIGIBILITY:
Inclusion Criteria:

1. Between 14 and 19 years of age upon entry into t-CARE
2. A primary diagnosis of Asperger's Syndrome or autism, as indicated by the Social Responsiveness Scale, Second Edition (SRS-2; Constantino & Gruber, 2012)
3. English as primary language spoken
4. Ability to self-report (i.e. understand and answer assessment questions written at a third grade comprehension level) (self-report questions to be asked by study coordinator)

Exclusion Criteria:

1. A significant language delay
2. Significant psychosis as indicated through a semi-structured interview (Mini-International Neuropsychiatric Interview)

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2016-01; Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Holmes and Rahe Stress Scale | annually over 2 years
SRS-2 | annually over 2 years
Waisman Activities of Daily Living Scale | annually over 2 years
Intolerance of Uncertainty | annually over 2 years
PROMIS Multi-Domain 49 | monthly over 2 years
Temple University Community Participation (TUCP) measure | quarterly over 2 years
PROMIS proxy measures | quarterly over 2 years
PROMIS SF measures | monthly over 2 years
Self-Determination Scale | annually over 2 years

SECONDARY OUTCOMES:
Closure Survey | after completion of 2 year study

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Murray, M.D., Principal Investigator — Hershey Medical Center
Locations (1):
- The Penn State College of Medicine, Hershey, Pennsylvania, United States